CLINICAL TRIAL: NCT07108985
Title: Prospective, Open-label, Randomized, Parallel-group, Multicenter, Investigator, Initiated Phase 4 Clinical Trial to Evaluate the Glycemic Lowering Effects of Adding SGLT2 Inhibitor Monotherapy, TZD Monotherapy, or SGLT2 Inhibitor/TZD Combination Therapy in Patients With Type 2 Diabetes on DPP4 Inhibitors
Brief Title: Effect of Add-on SGLT2i, TZD, or Combination Therapy in Type 2 Diabetes Patients on DPP4 Inhibitors
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2025-0720
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Hyperglycemia; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Insulin Resistance | interventions — Sitagliptin Phosphate; dapagliflozin; lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (Experimental): Sitagliptin 100 mg
  Interventions: Drug: Sitagliptin 100 mg
- B (Experimental): Sitagliptin 100 mg + Dapagliflozin 10 mg
  Interventions: Drug: Sitagliptin 100 mg + Dapagliflozin 10 mg
- C (Experimental): Sitagliptin 100 mg + Lobeglitazone 0.5 mg
  Interventions: Drug: Sitagliptin 100 mg + Dapagliflozin 10 mg
- D (Experimental): Sitagliptin 100 mg + Dapagliflozin 10 mg + Lobeglitazone 0.5 mg
  Interventions: Drug: Sitagliptin 100 mg + Dapagliflozin 10 mg + Lobeglitazone 0.5 mg

INTERVENTIONS:
Drug: Sitagliptin 100 mg — Sitagliptin 100 mg, taken once daily for 24 weeks.
  Arms: A
Drug: Sitagliptin 100 mg + Dapagliflozin 10 mg — Sitagliptin 100 mg + Dapagliflozin 10 mg, taken once daily for 24 weeks.
  Arms: B
Drug: Sitagliptin 100 mg + Dapagliflozin 10 mg — Sitagliptin 100 mg + Dapagliflozin 10 mg, taken once daily for 24 weeks.
  Arms: C
Drug: Sitagliptin 100 mg + Dapagliflozin 10 mg + Lobeglitazone 0.5 mg — Sitagliptin 100 mg + Dapagliflozin 10 mg + Lobeglitazone 0.5 mg, taken once daily for 24 weeks.
  Arms: D

SUMMARY:
This clinical trial investigates the effects of adding different diabetes medications to patients with type 2 diabetes who are currently being treated with DPP4 inhibitors. The study evaluates three treatment strategies: SGLT2 inhibitor monotherapy, TZD monotherapy, and a combination of both SGLT2 inhibitor and TZD. Participants will be randomly assigned to one of four groups, including a control group continuing DPP4 inhibitor alone.

The primary objective is to assess changes in blood sugar control, specifically HbA1c levels, after 12 and 24 weeks of treatment. Secondary outcomes include changes in fasting and postprandial glucose, insulin, C-peptide, lipid profiles (total cholesterol, triglycerides, HDL-C, LDL-C), body composition (muscle mass, visceral fat, subcutaneous fat), and insulin resistance indicators such as HOMA-IR, HOMA-beta, and Insulinogenic Index.

Eligible participants are adults aged 19 to 75 years with type 2 diabetes who have been on stable doses of DPP4 inhibitors, with or without metformin or sulfonylurea, for at least 8 weeks. Individuals with recent use of SGLT2 inhibitors or TZDs, significant organ dysfunction, or other exclusion criteria will not be enrolled.

The study is open-label and multicenter, conducted at four hospitals in Korea. All medications used in the trial are provided by the sponsor. Participants will receive lifestyle counseling throughout the study period, including guidance on diet and exercise. Safety monitoring will be conducted regularly, and adverse events will be documented and managed according to protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 19 and 75 years at the time of providing written informed consent.
2. Diagnosed with type 2 diabetes mellitus and having an HbA1c level between 7.5% and 11.0%.
3. Receiving DPP4 inhibitor monotherapy or combination therapy with metformin and/or sulfonylurea for at least 8 weeks without dose adjustment.
4. Provided written informed consent voluntarily after receiving a full explanation of the study.
5. Considered capable of understanding the study procedures and cooperating throughout the study period until completion.

Exclusion Criteria:

1. Patients with diabetes other than type 2 diabetes, including type 1 diabetes or gestational diabetes.
2. Use of TZD or SGLT2 inhibitors within the past 8 weeks, or history of discontinuation due to serious adverse reactions.
3. Currently receiving four or more antidiabetic medications.
4. History of diabetic ketoacidosis (with or without coma) or acute/chronic metabolic acidosis within the past 24 weeks.
5. Known allergy or hypersensitivity to the investigational drugs or their components.
6. Chronic use (more than 14 consecutive days) of oral or parenteral corticosteroids within 8 weeks prior to screening, with ongoing need for dose adjustment.
7. Genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
8. Active or progressive malignant tumors requiring treatment.
9. History of drug abuse or alcohol dependence within the past 12 weeks.
10. HIV infection.
11. Severe infections, perioperative status, or major trauma.
12. History of heart failure classified as NYHA class III or IV within the past 24 weeks.
13. History of acute cardiovascular events within the past 12 weeks (e.g., unstable angina, myocardial infarction, transient ischemic attack, stroke, coronary artery bypass grafting, or coronary intervention).
14. Renal failure or chronic kidney disease with eGFR < 25 mL/min/1.73m² or undergoing dialysis.
15. Active bladder cancer or history of bladder cancer.
16. Abnormal liver function defined as serum ALT, AST, or alkaline phosphatase > 5× ULN, or total bilirubin > 5× ULN.
17. Pregnant or breastfeeding women.
18. Participation in another clinical trial or administration of investigational drugs within the past 12 weeks (except for observational or retrospective studies deemed not to affect the safety or efficacy of this trial).
19. Determined by the investigator to be unsuitable for participation in the study.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
change in HbA1c levels | At 12 and 24 weeks after initiation of the investigational drug
  To assess the change in HbA1c levels at 12 and 24 weeks after administration of the investigational drugs, by comparing pre- and post-treatment values within each group and between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, 50-1 Yonsei-ro, Seodaemun-gu, Seoul 03722, Republic of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No